CLINICAL TRIAL: NCT06907680
Title: A Randomized Placebo-controlled Crossover Trial Assessing the Efficacy and Safety of M-Gard Particulate EW in the Treatment of Seasonal Allergic Rhinitis
Brief Title: M-Gard Particulate EW Efficacy Study on Seasonal Allergic Rhinitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: RDC Clinical Pty Ltd (Industry)
Collaborators: Lallemand Bio-Ingredients (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BETALL
Record Dates: First submitted 2025-03-27; First posted 2025-04-02 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-03

CONDITIONS: Allergic Rhinitis Due to Grass Pollens
Keywords: allergic rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, cross-over trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- M-Gard (Experimental): One capsule containing 250mg of M-Gard Particulate EW is taken twice daily for 14 days.
  Interventions: Dietary Supplement: M-Gard
- Placebo (Placebo Comparator): One capsule containing 250mg of MCC (Microcrystalline Cellulose) is taken twice daily for 14 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: M-Gard — One capsule containing 250mg of M-Gard Particulate EW is taken twice daily for 14 days.
  Other Names: M-Gard Particulate EW
  Arms: M-Gard
Other: Placebo — One capsule containing 250mg of MCC (Microcrystalline Cellulose) is taken twice daily for 14 days.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to assess the efficacy and safety of M-Gard supplementation for alleviating the symptoms of allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years.
* Generally healthy
* Individuals with a history of recurrent seasonal allergic rhinitis
* Positive RAST test for grass allergy
* BMI 18-35kg/m2
* Able to provide informed consent
* Agree not to change current diet and/or exercise routine during entire enrolment period
* Agree to not participate in another clinical trial during the study period

Exclusion Criteria:

* Serious illness e.g., liver disease, kidney disease, heart disease, mood disorders, neurological disorders such as multiple sclerosis.
* Unstable illness e.g., diabetes and thyroid gland dysfunction.
* Current malignancy (excluding Basal Cell Carcinoma) or chemotherapy or radiotherapy treatment for malignancy within the previous 2 years.
* Individuals with symptomatic perennial allergic rhinitis, non-allergic rhinitis, chronic respiratory conditions (e.g., asthma, chronic obstructive pulmonary disease).
* Participants with cognitive damage.
* Acute illness experienced in the past 1 month.
* Active smokers and/or nicotine or drug abuse.
* Allergic to any of the ingredients in the active or placebo formula.
* Chronic past and/or current alcohol use (>21 alcoholic drinks per week)
* Attempting to conceive, pregnant or lactating women
* Use of medications that would affect the immune and/or the inflammatory response e.g. immunotherapy, antihistamines (daily use), corticosteroids, mast cell stabilizers, leukotriene modifiers, and decongestants.
* Currently taking Coumadin (Warfarin), Heparin, Dalteparin, Enoxaparin or other anticoagulation therapy including low dose aspirin; tricyclic antidepressants; Clonidine and other central acting alpha-2-agonists.
* Participants who are currently participating in any other clinical trial or who have participated in any other clinical trial during the past 1 month.
* Any condition which in the opinion of the investigator makes the participant unsuitable for inclusion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Relief of symptoms of allergic rhinitis | Day 0 to Day 43
  Relief of symptoms of allergic rhinitis, as measured by:
  Total and individual allergic rhinitis symptom severity as measured by a visual analogue scale (VAS) of nasal congestion, sneezing, itchy nose, runny nose and watery eyes. These symptoms will be rated on a scale of 0 to 10 where 0 is "not troublesome at all" and 10 is "very troublesome".

SECONDARY OUTCOMES:
Reflective Total Nasal Symptom Scores (rTNSS) | Day 0 to Day 43
  Change from baseline to the end of the study period in Reflective Total Nasal Symptom Scores (rTNSS). Self-reported questionnaire rating the severity of four nasal symptoms (runny nose, nasal congestion, itchy nose, and sneezing) on a four-point scale (0-3), where 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms, and 3 = severe symptoms. The rTNSS is the sum of the scores for each of the nasal symptoms (from 0 to 12)
Reflective Total Ocular Symptom Scores (rTOSS) | Day 0 to Day 43
  Change from baseline to the end of the study period in Reflective Total Ocular Symptom Scores (rTOSS). Self-reported questionnaire that is calculated as the sum of the patients' scoring of the severity of three ocular symptoms (itching/burning, tearing/watering, and redness) on a scale of 0-3 where 0 = absent, 1 = mild, 2 = moderate, and 3 = severe).
Rhinitis Control Scoring System (RCSS) | Day 0 to Day 43
  Change from baseline to the end of the study period in Rhinitis Control Scoring System (RCSS). Subject-completed tool including 5 items (sneezing, rhinorrhoea, nasal obstruction, nasal pruritus, and conjunctivitis). Each symptom is rated on a 5-point scale depending on its intensity (none-10%, mild-8%, moderate-6%, severe-4%, very severe-2%) and its frequency (never-10%, rarely-8%, occasionally-6%, frequently-4%, very frequently-2%), which are assessed separately. The sum of the intensity score and the frequency score gives the global score
Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ). | Day 0 to Day 43
  Change from baseline to the end of the study period in Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ). Self-reported questionnaire used measure the functional impairments that are most troublesome to patients because of their rhinoconjunctivitis. It consists of 28 questions in 7 domains (activity limitation, sleep problems, nose symptoms, eye symptoms, non-nose/eye symptoms, practical problems and emotional function). These are rated on a 7-point scale (0 = not impaired at all - 6 = severely impaired).
Peak Nasal Inspiratory Flow (PNIF) | Day 0 to Day 43
  Change from baseline to the end of the study period in Peak Nasal Inspiratory Flow (PNIF). Peak nasal inspiratory flow (PNIF) is a measure of nasal patency and measures the maximum airflow a patient is able to produce during forced nasal inspiration. PNIF (in L/min) will be measured with a peak inspiratory flow meter. The highest of three successive measurement values will be recorded
Onset of action of treatment | Day 12 and Day 41
  Change from baseline to the end of the study period in onset of action of treatment, this will be measured during the nasal allergen challenge. Peak nasal inspiratory flow (PNIF) will be measured to assess for nasal patency and allergy symptoms will be rated via the VAS, rTNSS, rTOSS, RCSS and RQLQ.
  The time from the onset of symptoms to their resolution will be measured.
Pathology markers | Day 0 to Day 41
  Change from baseline to the end of the study period in Pathology markers: cytokines, histamine, tryptase, allergen specific IgE.
Use of rescue /concomitant medications | Day 0 to Day 43
  Change from baseline to the end of the study period in use of rescue /concomitant medications.
Safety - Adverse events | Day 0 to Day 43
  Change from baseline to the end of the study period in Safety via Adverse Event reporting and incident rate ratio between placebo and treatment groups.
Safety - Vital Signs (Blood Pressure) | Day 0 to Day 41
  Change from baseline to the end of the study period in Safety via Vital Signs (blood pressure).
Safety - Vital Signs (Heart Rate) | Day 0 to Day 41
  Change from baseline to the end of the study period in Safety via Vital Signs heart rate.
Safety - Vital Signs (O2 saturation) | Day 0 to Day 41
  Change from baseline to the end of the study period in Safety via Vital Signs (O2 saturation).
Safety - Vital Signs (temperature) | Day 0 to Day 41
  Change from baseline to the end of the study period in Safety via Vital Signs (temperature).
Safety - Safety Markers (FBC) | Day 0 to Day 41
  Change from baseline to the end of the study period in Safety via Safety Markers (Full Blood Count).
Safety - Safety Markers (E/LFT) | Day 0 to Day 41
  Change from baseline to the end of the study period in Safety via Safety Markers (E/LFT).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Tompkins, Study Director — Lallemand Bio-Ingredients
Locations (1):
- RDC Clinical, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: Undecided